CLINICAL TRIAL: NCT02347384
Title: A Prospective, Randomized, Multicenter Clinical Study in Chinese Subjects to Compare the Safety and Efficacy of the Delta PLUS Femoral Head and SL-TWIN Stem With BIOLOX Forte Ball Head and SL-PLUS Stem in Total Hip Arthroplasty
Brief Title: Project JAY THA Registration Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Smith & Nephew Orthopaedics (Beijing) Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-4560-02
Record Dates: First submitted 2015-01-09; First posted 2015-01-27 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis; Post-traumatic Arthritis; Avascular Necrosis; Developmental Dysplasia of the Hip; Femoral Neck Fracture
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Osteonecrosis; Developmental Dysplasia of the Hip; Femoral Neck Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Delta PLUS Femoral Head + SL-TWIN Stem (Experimental): Subject will be implanted with Delta PLUS Femoral Head & SL-TWIN Stem
  Interventions: Device: Delta PLUS Femoral Head + SL-TWIN Stem
- BIOLOX forte ball head + SL-PLUS Stem (Active Comparator): Subject will be implanted with BIOLOX forte ball head & SL-PLUS Stem
  Interventions: Device: BIOLOX forte ball head + SL-PLUS Stem

INTERVENTIONS:
Device: Delta PLUS Femoral Head + SL-TWIN Stem — Subject will undergo total hip arthroplasty with Delta PLUS Femoral Head & SL-TWIN Stem
  Arms: Delta PLUS Femoral Head + SL-TWIN Stem
Device: BIOLOX forte ball head + SL-PLUS Stem — Subject will undergo total hip arthroplasty with BIOLOX forte ball head & SL-PLUS Stem
  Arms: BIOLOX forte ball head + SL-PLUS Stem

SUMMARY:
This is a prospective, randomized, multicenter clinical study in Chinese subjects to compare the safety and efficacy of the Delta PLUS Femoral Head and SL-TWIN Stem with BIOLOX forte ball head and SL-PLUS Stem in total hip arthroplasty

DETAILED DESCRIPTION:
As the incidence of joint disease continues to increase, an ever growing percentage of the affected population will undergo total hip arthroplasty (THA). This recent upward trend for THA procedures appears to be directly related to the prevalence of certain health factors. Specifically, longer life spans, rising obesity rates, and increasing physical activity levels in relatively younger populations are all examples of factors that may significantly contribute to hip degeneration. While strategies such as weight reduction, lifestyle change, or drug therapy may offer temporary relief from the symptoms of joint degeneration, THA remains the standard of care for subjects experiencing significant losses in quality of life due to advanced hip disease.

There has been an increase in imported hip prostheses during the past decade, so that surgeons now have more choices of implants. However, the high cost of imported prostheses has become a barrier to the development of hip replacement in China and caused many patients requiring immediate hip replacement to have to delay or miss their surgery. The development and promotion of high-quality domestic joint implants and surgical instruments is the key to the development of joint replacement technique in China.

The primary objective of this study is to demonstrate non-inferiority of subjects implanted with the Delta PLUS Femoral Head + SL-TWIN Stem compared to a randomized concurrent control group of subjects implanted with the BIOLOX forte ball head + SL-PLUS Stem in terms of mean Harris Hip Score (HHS) at 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, aged between 50 and 75 years inclusive of Chinese ethnicity.
* Subject presents with osteoarthritis, rheumatoid arthritis, post-traumatic arthritis, avascular necrosis of hip joint, developmental dysplasia of the hip, or femoral neck fracture requiring primary total hip replacement.
* Subject who is able to give voluntary, written informed consent to participate in the study and from whom consent has been obtained by signing and dating an EC-approved consent form.
* Subject who is able to understand this clinical study, co-operates with the investigational procedures and is willing to return to the hospital for all the required post-operative follow-ups for up to 12 months.
* Life expectancy of subject is over 2 years.

Exclusion Criteria:

* Bilateral hip disease with the anticipated need for bilateral hip implant during study participation (i.e., within the next 12 months).
* Subject experienced prior joint replacement surgery on any major joint (hip, knee) in lower limb within the last 12 months.
* Subject with developmental dysplasia of the hip of CROWE grade 3 or 4.
* Subject has known or suspected metal sensitivity.
* Subject is known to have insufficient bone stock resulting from conditions such as cancer, significant osteoporosis or metabolic bone disorders, which cannot provide adequate support and/or fixation to the prosthesis.
* Subject is severely obese (BMI>35).
* Subject had an active infection or sepsis (treated or untreated).
* Subject has conditions that may compromise implant stability or postoperative recovery (i.e., Paget's or Charcot's disease, vascular insufficiency, muscular atrophy, uncontrolled diabetes, moderate to severe renal insufficiency, hip abduction muscle strength less than grade IV or complete loss, or neuromuscular disease).
* Subject has an emotional or neurological condition that would affect their ability or willingness to participate in the study (e.g. cognitive disorder, mental illness, mental retardation).
* Subject is immunosuppressed, has an autoimmune disorder, or an immunosuppressive disorder. For examples, subject is on immunosuppressive therapy (corticosteroid hormones in large amounts, cytotoxic drugs, antilymphocytic serum or irradiation in large doses) or has acquired immunodeficiency syndrome (AIDS).
* Subject is known to be at risk for lost to follow-up, or failure to return for scheduled visits.
* Subject was enrolled in another investigational drug, biologic, or device study in the last 12 months.
* Subject is a woman who is pregnant or lactating，or intends to become pregnant during the course of the study.
* Known alcohol and/or drug abuse

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-04-20; Primary Completion 2016-11-01 (Actual); Study Completion 2016-11-01 (Actual)

PRIMARY OUTCOMES:
Harris Hip Score | 1 year post-operative

SECONDARY OUTCOMES:
Composite Clinical Success, as indicated by A) No revision of any device component; and B) Total Harris Hip Score greater than or equal to 80 (excellent to good score); and C) Radiologic success. | 1 year post-operative
  A successful individual outcome for a subject in total hip arthroplasty will be characterized at 1 year postoperative by a composite of three success criteria:
  A. No revision of any device component; and B. Total Harris Hip Score greater than or equal to 80 (excellent to good score); and C. Radiologic success.

OTHER OUTCOMES:
The Western Ontario and McMaster Universities Arthritis Index(WOMAC) | 1 year post-operative
SF-12 Health Survey | 1 year post-operative
Number of adverse events | Up to 1 year post-operative

CONTACTS AND LOCATIONS:
Overall Officials: Li Cao, Study Chair — First Affiliated Hospital of Xinjiang Medical University
Locations (4):
- China (4):
  - Luoyang Orthopedic-Traumatological Hospital, Luoyang, Henan
  - Inner Mongolia Bao Gang Hospital, Baotou, Inner Mongolia
  - The First Teaching Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Traditional Chinese Medicine Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang

IPD SHARING:
Plan to Share IPD: No